CLINICAL TRIAL: NCT07046416
Title: Effectiveness of Occupation-Based Exercise Program Added to Conventional Rehabilitation Program on Hand Functions, Range of Motion, Grip Strength, Pain and Kinesiophobia in Zone 2 Flexor Tendon Injuries
Brief Title: Effectiveness of Occupation-Based Exercise Program in Zone 2 Flexor Tendon Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berat Güngör (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor-Investigator, Berat Güngör, Dr., Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3005950
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Tendon Injuries; Zone 2 Flexor Tendon Lacerations of the Hand
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupation-based exercise group (Experimental)
  Interventions: Other: Occupation-Based Exercise Program
- Conventional therapy group (Active Comparator)
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: Occupation-Based Exercise Program — In the occupation-based exercise program, while trying to improve the range of motion and muscle strength of the hand, it is aimed to successfully return to daily life activities. For this reason daily activities are used instead of memorized range movements. In this way, the occupation-based exercise program provides a physical recovery in patients with hand injuries, while providing positive improvements in parameters related to the mind and spirit. Patients' participation, motivation and compliance with the treatment are increased in the hand rehabilitation process, which can be challenging for patients.
  In addition to the conventional treatment program, the study/experimental group, will be given occupation-based exercises for a total of 4 weeks between the 6th and 10th weeks postoperatively, 2 days a week with a physiotherapist and the other days with a home program.
  Arms: Occupation-based exercise group
Other: Conventional therapy group — Conventional group treatment will be according the early passive hand rehabilitation program. Conventional group will be followed with a cast-splint made by the surgical team for the first 4 weeks within the scope of the conventional treatment program. From the 4th week onwards, the duration of splint use is gradually reduced and is completely discontinued from the 6th week onwards. At the end of the 4th week, depending on the wound condition, contrast bath, scar massage, retrograde massage, active and passive flexion, active extension and tendon shifting exercises are applied as tolerated. After the 6th week, isolated block exercises and stretching exercises are added if there is contracture. Strengthening exercises are started from the 8th-10th week.
  Arms: Conventional therapy group

SUMMARY:
Aim of the study is to evaluate the effects of a 4-week occupation-based exercise program given in addition to the conventional rehabilitation program on hand functions, range of motion, grip strength, pain and kinesiophobia in the post-operative rehabilitation of patients aged 18-65 years with zone 2 flexor tendon repair.

Expected results: To prove the effectiveness of occupation-based exercises in order to reduce the failure rates seen in the rehabilitation of zone 2 flexor tendon injuries, to increase patient compliance and motivation during the rehabilitation process, to improve functional outcomes by ensuring its inclusion in conventional treatment and to increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Flexor zone 2 injury
* At least 1 flexor digitorum superfisialis or flexor digitorum profundus tendon repair
* No visual and hearing impairment
* Have the cognitive function to coordinate and carry out simple commands

Exclusion Criteria:

* Concomitant flexor pollicis longus tendon injury
* Concomitant extensor tendon injury
* Accompanying fracture
* Associated median/ulnar/radial nerve injury
* Less than 50% partial flexor tendon injury
* Cognitive impairment resulting in an inability to understand and carry out simple commands
* Not being able to comply with the rehabilitation protocol to be applied after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disabilities of The Arm, Shoulder and Hand Questionnaire (DASH) | Participants will be evaluated at 6th, 10th and 16th weeks postoperative.
  In DASH Questionnaire a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score on both test ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
Modified Strickland Classification | Participants will be evaluated at 6th, 10th and 16th weeks postoperatively.
  Range of motion of the fingers will be measured with a goniometer and results will classified according to Modified Strickland Classification
Numerical Pain Rating Scale (NPRS) | Participants will be evaluated at 6th, 10th and 16th weeks postoperatively.
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Tampa Kinesiophobia Scale | Participants will be evaluated at 6th, 10th and 16th weeks postoperatively
  The scale total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Grip strentgh | Participants will be evaluated at 6th, 10th and 16th weeks postoperatively.
  Hand grip strength will be measured with a hand dynamometer and finger grip strength with a pinchmeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıversity, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)